CLINICAL TRIAL: NCT03804931
Title: Efficacy and Safety of Fecal Microbiota Transplantation for Ulcerative Colitis
Brief Title: Fecal Microbiota Transplantation for Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K-2017-103-01
Record Dates: First submitted 2019-01-06; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-11

CONDITIONS: Ulcerative Colitis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Prednisone; Mesalamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fecal microbiota transplantation (Experimental): Fecal microbiota transplantation
  Interventions: Procedure: Fecal microbiota transplantation; Drug: 5-Aminosalicylic acid(5-ASA) and/or Prednisone
- placebo fecal microbiota transplantation (Sham Comparator): Infusion of Saline
  Interventions: Procedure: Infusion of Saline; Drug: 5-Aminosalicylic acid(5-ASA) and/or Prednisone
- Traditional treatments (Other): Drug:5-Aminosalicylic acid(5-ASA) and/or Prednisone
  Interventions: Drug: 5-Aminosalicylic acid(5-ASA) and/or Prednisone

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — 200 mL of prepared fecal microbiota suspension from healthy donors' fresh feces was injected into the intestine
  Arms: Fecal microbiota transplantation
Procedure: Infusion of Saline — Infusion of Saline
  Arms: placebo fecal microbiota transplantation
Drug: 5-Aminosalicylic acid(5-ASA) and/or Prednisone — Mesalazine and/or Prednisone
  Other Names: Mesalazine; Prednisone

SUMMARY:
Fecal microbiota transplantation (FMT) is a strategy that infuses a fecal suspension containing a healthy donor's microbiota into a patient's gut to restore his/her intestinal microbiome. Fecal microbiota transplantation has been used for several disease，but the efficacy of ulcerative colitis(UC) by fecal microbiota transplantation needs to be further explored.The investigators propose to determine the efficiency and safety of FMT in patients with ulcerative colitis(UC).

DETAILED DESCRIPTION:
The present clinical trial aims to re-establish a gut functionality state of intestinal flora through FMT as a therapy for ulcerative colitis(UC). We established a standard microbiota isolation from donated fresh stool in lab. Then the microbiota is transplanted to the intestine. Patients from Guangzhou First People's Hospital in this study will be assigned to receive FMT at least two times according to associated guidelines and follow-up for at least three months.

ELIGIBILITY:
Inclusion Criteria:

* Active, moderate to severe severity (Mayo score more than 6)
* Safety using history of 5-ASA
* Able to undergo endoscopy examination

Exclusion Criteria:

* Antibiotic using in 7 days
* High risk of toxic megacolon
* Colon cancer or neoplasia in pathophysiology
* Other severe diseases (eg: cardiovascular, respiratory, gastroenteral and kidney diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission in patient as assessed using Mayo score | 12 weeks
  Total Mayo score less than 2 and no signal item more than 1
Clinical improvement in patient as assessed using Mayo score | 12 weeks
  Total Mayo score decreased more than 3

SECONDARY OUTCOMES:
Intestinal microbiota changing | 12 weeks
  The change of intestinal microbiota composition after FMT compared with subject original microbiota and donor's microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Yuqiang Nie, MD, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui B, Li P, Xu L, Zhao Y, Wang H, Peng Z, Xu H, Xiang J, He Z, Zhang T, Nie Y, Wu K, Fan D, Ji G, Zhang F. Step-up fecal microbiota transplantation strategy: a pilot study for steroid-dependent ulcerative colitis. J Transl Med. 2015 Sep 12;13:298. doi: 10.1186/s12967-015-0646-2. PMID 26363929